CLINICAL TRIAL: NCT01562158
Title: A Multi-centre, Randomised, Double-blind, Parallel Groups, Placebocontrolled Trial on Efficacy and Safety of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in Treatment of Bleeding in Patients Following Stem Cell Transplantation (SCT)
Brief Title: Efficacy and Safety of Activated Recombinant Human Factor VII in Treatment of Bleeding in Patients Following Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7BMT-1360
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Bleeding During/Following Surgery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Procedure: standard therapy; Drug: placebo
- Low dose (Experimental)
  Interventions: Procedure: standard therapy; Drug: activated recombinant human factor VII
- Medium dose (Experimental)
  Interventions: Procedure: standard therapy; Drug: activated recombinant human factor VII
- High dose (Experimental)
  Interventions: Procedure: standard therapy; Drug: activated recombinant human factor VII

INTERVENTIONS:
Procedure: standard therapy — Standard treatment of bleeding
Drug: activated recombinant human factor VII — Two days repeated treatment regimen - low dose administered i.v. (into the vein)
  Arms: Low dose
Drug: activated recombinant human factor VII — Two days repeated treatment regimen - medium dose administered i.v. (into the vein)
  Arms: Medium dose
Drug: activated recombinant human factor VII — Two days repeated treatment regimen - high dose administered i.v. (into the vein)
  Arms: High dose
Drug: placebo — Placebo
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia, Europe and Oceania. The aim of this trial is to evaluate the efficacy of placebo and activated recombinant human factor VII in patients having undergone allogeneic or autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone allogeneic or autologous stem cell transplantation

Exclusion Criteria:

* Known or suspected allergy to trial product
* Participation in other trials with unapproved drugs or trials with equal or similar objective

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-04; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Effect on bleeding, defined as change in bleeding score

SECONDARY OUTCOMES:
Transfusion requirements
Bleeding evaluation
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (43):
- Novo Nordisk Investigational Site, Chapel Hill, North Carolina, United States
- Australia (3):
  - Novo Nordisk Investigational Site, Herston
  - Novo Nordisk Investigational Site, Parkville
  - Novo Nordisk Investigational Site, Westmead
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Copenhagen, Denmark
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (3):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Tours
- Germany (9):
  - Novo Nordisk Investigational Site, Cologne
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Idar-Oberstein
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Regensburg
  - Novo Nordisk Investigational Site, Tübingen
  - Novo Nordisk Investigational Site, Wiesbaden
- Israel (2):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
- Italy (5):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Pesaro
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Udine
- Poland (5):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, Singapore, Singapore
- Spain (3):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Valencia
- Sweden (3):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Uppsala
- Switzerland (2):
  - Novo Nordisk Investigational Site, Basel
  - Novo Nordisk Investigational Site, Zurich
- Novo Nordisk Investigational Site, Bangkok, Thailand
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Result] Pihusch M, Bacigalupo A, Szer J, von Depka Prondzinski M, Gaspar-Blaudschun B, Hyveled L, Brenner B; F7BMT-1360 Trial Investigators. Recombinant activated factor VII in treatment of bleeding complications following hematopoietic stem cell transplantation. J Thromb Haemost. 2005 Sep;3(9):1935-44. doi: 10.1111/j.1538-7836.2005.01523.x. PMID 16102099
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com